CLINICAL TRIAL: NCT06100172
Title: Delivering Transcutaneous Auricular Neurostimulation as an Adjunct Non-Opioid Pain Management Therapy for Patients Undergoing Lumbar Surgery
Brief Title: Transcutaneous Auricular Neurostimulation After Lumbar Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Alex Valadka, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU-2023-0197
Record Dates: First submitted 2023-09-14; First posted 2023-10-25 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Pain, Postoperative; Opioid Use; Lumbar Spine Injury
Keywords: Lumbar Surgery; Transcutaneous auricular neurostimulation (tAN)
MeSH Terms: conditions — Pain, Postoperative; Spinal Injuries

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, sham controlled.
Who Masked: Participant, Investigator
Masking Description: On the day of surgery, subjects will be randomized 1:1 to either the active stimulation group or the sham group. In the sham group, the device looks like the active device, but it will not deliver any electrical stimulation to the vagus or trigeminal nerves.
  Both groups will receive the SOC for post-operative pain management for lumbar surgery patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active tAN + standard of care (SOC) for post-operative pain management for lumbar spine patients. (Active Comparator): Subjects will be randomized to receive the active device on the day of surgery.
  Subjects will receive treatment according to the following time points:
  * Pre-operative: 30 minutes in the hour prior to surgery
  * Intra-operative: 30 minutes before the end of surgery
  * Post-operative: 30 minutes at 3 and 6 hours after surgery
  * Inpatient: Four 30-minute sessions on Day 2
  Interventions: Device: Sparrow Ascent Transcutaneous Auricular Neurostimulation (tAN)
- Sham tAN + standard of care (SOC) for post-operative pain management for lumbar spine patients. (Placebo Comparator): Subjects will be randomized to receive the sham device on the day of surgery.
  Subjects will receive treatment according to the following time points:
  * Pre-operative: 30 minutes in the hour prior to surgery
  * Intra-operative: 30 minutes before the end of surgery
  * Post-operative: 30 minutes at 3 and 6 hours after surgery
  * Inpatient: Four 30-minute sessions on Day 2
  Interventions: Device: Sham Control Device

INTERVENTIONS:
Device: Sparrow Ascent Transcutaneous Auricular Neurostimulation (tAN) — This method of simultaneous vagal and trigeminal stimulation via the external ear is known as transcutaneous auricular neurostimulation (tAN), as the targets of electrical stimulation include the auricular branch of the vagus nerve (ABVN) and auriculotemporal nerve (ATN), which is a branch of the mandibular division of the trigeminal nerve. Electrodes applied to select dermatome regions can target ear neural structures and deliver non-invasive vagus nerve stimulation (VNS) and trigeminal nerve stimulation (TNS). Use of tAN for pain relief is an attractive alternative to pharmacologic and opioid-based approaches because it is safe and effective and presents no addiction liability.
  Arms: Active tAN + standard of care (SOC) for post-operative pain management for lumbar spine patients.
Device: Sham Control Device — This device looks like the active device, but no stimulation will be delivered.
  Arms: Sham tAN + standard of care (SOC) for post-operative pain management for lumbar spine patients.

SUMMARY:
The purpose of this study, entitled "Delivering Transcutaneous Auricular Neurostimulation as an Adjunct Non-Opioid Pain Management Therapy for Patients Undergoing Lumbar Surgery", is to demonstrate whether transcutaneous auricular neurostimulation (tAN) can non-invasively reduce the perception of pain in patients undergoing lumbar surgery. tAN is placed on and around the ear to non-invasively stimulate branches of the vagus and trigeminal nerves and modulate specific brain regions associated with pain.

DETAILED DESCRIPTION:
This study is designed as a randomized, double-blind, sham-controlled, single-center, clinical trial in which 20 patients undergoing lumbar spine surgery will be randomized 1:1 into one of two treatment groups:

1. Group 1 (n=10): Active tAN + standard care
2. Group 2 (n=10): Sham tAN + standard care

Stimulation:

Participants undergoing lumbar surgery will be randomized to receive either active or sham tAN treatment according to the following time points:

* Pre-operative: 30 minutes in the hour prior to surgery
* Intra-operative: 30 minutes before the end of surgery
* Post-operative: 30 minutes at 3 and 6 hours after surgery
* Inpatient: Four 30-minute sessions on Day 2

Blood Draws

Participants will have blood samples collected at the following time points:

* Day 1 (Day of Surgery)
* Day 2 (Day 1 post-surgical)

Follow up Visits Participants will have study follow up visits on Days 7 and Day 14. These visits can either be conducted either via a secure telehealth video visit, or in person visit.

ELIGIBILITY:
Inclusion Criteria:

1. Medically cleared to undergo a lumbar spine surgery, either spinal fusion with or without multilevel laminectomies, or lumbar multilevel laminectomies alone.
2. 18-85 years of age
3. English Proficiency
4. Participants must be able to provide informed consent and function at an intellectual level sufficient for study requirements

Exclusion Criteria:

1. Current evidence of an uncontrolled and/or clinically significant medical condition
2. History of bleeding disorders or coagulopathy
3. History of seizures or epilepsy
4. History of neurological diseases or traumatic brain injury
5. Use of illegal recreational drugs
6. Presence of devices, e.g. pacemakers, cochlear prosthesis, neuro-stimulators
7. Use of acupuncture within 4 weeks of surgery
8. Grossly abnormal external ear anatomy or active ear infection
9. Women of childbearing potential, not using effective contraception per investigator judgment or not willing to comply with contraception for the duration of the study
10. Females who are pregnant or lactating
11. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Pain Scores on the Visual Analog Scale (VAS) at 3 hours post-operation | Baseline, 3 hours post-operation
  Patients will be asked to report their level of pain using the Visual Analog Scale. Possible scores for VAS pain scale ranges from 0-10 where 0="no pain" to 10="severe pain"
Change From Baseline in Pain Scores on the Visual Analog Scale (VAS) at 6 hours post-operation | Baseline, 6 hours post-operation
  Patients will be asked to report their level of pain using the Visual Analog Scale. Possible scores for VAS pain scale ranges from 0-10 where 0="no pain" to 10="severe pain"
Change From Baseline in Pain Scores on the Visual Analog Scale (VAS) at day 2 post-operation | Baseline, day 2 post-operation
  Patients will be asked to report their level of pain using the Visual Analog Scale. Possible scores for VAS pain scale ranges from 0-10 where 0="no pain" to 10="severe pain"
Change From Baseline in Pain Scores on the Visual Analog Scale (VAS) at day 14 post-operation | Baseline, day 14 post-operation
  Patients will be asked to report their level of pain using the Visual Analog Scale. Possible scores for VAS pain scale ranges from 0-10 where 0="no pain" to 10="severe pain"

SECONDARY OUTCOMES:
Mean total postoperative opioid consumption (morphine equivalent dose) at 3 hours post-surgery | 3 hours post-surgery
  During the in-patient hospital stay, the dose and frequency of post -operative opioid use will recorded for both the placebo and active groups. The opioid usage between the 2 groups will be compared to determine if the active group required less opioid medications for pain reduction.
Mean total postoperative opioid consumption (morphine equivalent dose) at 6 hours post-surgery | 6 hours post-surgery
  During the in-patient hospital stay, the dose and frequency of post -operative opioid use will recorded for both the placebo and active groups. The opioid usage between the 2 groups will be compared to determine if the active group required less opioid medications for pain reduction.
Mean total postoperative opioid consumption (morphine equivalent dose) at Day 2 post-surgery | Day 2 post-surgery
  During the in-patient hospital stay, the dose and frequency of post -operative opioid use will recorded for both the placebo and active groups. The opioid usage between the 2 groups will be compared to determine if the active group required less opioid medications for pain reduction.
Mean total postoperative opioid consumption (morphine equivalent dose) at Day 7 post-surgery | Day 7 post-surgery
  During the in-patient hospital stay, the dose and frequency of post -operative opioid use will recorded for both the placebo and active groups. The opioid usage between the 2 groups will be compared to determine if the active group required less opioid medications for pain reduction.
Mean total postoperative opioid consumption (morphine equivalent dose) at Day 14 post-surgery | Day 14 post-surgery
  During the in-patient hospital stay, the dose and frequency of post -operative opioid use will recorded for both the placebo and active groups. The opioid usage between the 2 groups will be compared to determine if the active group required less opioid medications for pain reduction.
Mean percent change in C-reactive protein (CRP) levels from baseline at Day 1 (intra-op) | Baseline and at Day 1 (intra-op)
  CRP blood samples collected will be used to measure the amount of inflammation in the body at the time points stated, and changes will be recorded and compared between the 2 groups. Plasma levels of C-reactive protein will be determined by the immunoprecipitation method using an in vitro diagnostic assay.
Mean percent change in C-reactive protein (CRP) levels from baseline at 6 hours post-op | Baseline and at 6 hours post-op
  CRP blood samples collected will be used to measure the amount of inflammation in the body at the time points stated, and changes will be recorded and compared between the 2 groups. Plasma levels of C-reactive protein will be determined by the immunoprecipitation method using an in vitro diagnostic assay.
Mean percent change in C-reactive protein (CRP) levels from baseline at Day 2 post-op | Baseline and at Day 2 post-op
  CRP blood samples collected will be used to measure the amount of inflammation in the body at the time points stated, and changes will be recorded and compared between the 2 groups. Plasma levels of C-reactive protein will be determined by the immunoprecipitation method using an in vitro diagnostic assay.
Mean percent change in Tumor Necrosis factor (TNF)-alpha levels from baseline at Day 1 (intra-op) | Baseline and at Day 1 (intra-op)
  TNF-alpha blood samples collected will be used to measure the amount of inflammation in the body at the time points stated, and changes will be recorded and compared between the 2 groups.
Mean percent change in TNF-alpha levels from baseline at 6 hours post-op | Baseline and at 6 hours post-op
  TNF-alpha blood samples collected will be used to measure the amount of inflammation in the body at the time points stated, and changes will be recorded and compared between the 2 groups.
Surgery time (incision to closure) | Day 1- during surgery [Surgery start (incision) to closure of surgical site]
  A comparison of the surgery times from incision to closure will be compared between the 2 groups to determine if the tAN affects the surgery time. The times will be recorded for each case, and then compared between the two groups. Surgery time - calculated as time from first incision to closure.
Estimated mean total blood loss | Day 1- During surgery [Surgery start (incision) to closure]
  During surgery, blood will be collected using cell saver technology which allows for accurate recording of total blood loss. The volume of blood loss will be recorded for each case, and then the 2 groups will be compared. Comparison is based on end volume recorded at incision closure.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Valadka, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No